CLINICAL TRIAL: NCT03486340
Title: Prevention of CArdioToxic-related CHest Pain in Cancer Patients Treated With 5-fluorouracil
Brief Title: Prevention of Chest Pain in Chemo-treated Cancer Patients
Acronym: CATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Collaborators: Region of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CATCH2018
Record Dates: First submitted 2018-03-26; First posted 2018-04-03 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Solid Carcinoma; 5-Fluorouracil Toxicity; Cardiotoxicity; Chemotherapeutic Toxicity; Acute Coronary Syndrome; Coronary Artery Calcification; Chest Pain
MeSH Terms: conditions — Cardiotoxicity; Acute Coronary Syndrome; Chest Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiological assessment (Experimental): a sub-acute cardiologic assessment and aggressive management of risk factors before oncologic treatment
  Interventions: Procedure: Cardiologic assessment
- Standard treatment (No Intervention): Standard chemotherapeutic treatment

INTERVENTIONS:
Procedure: Cardiologic assessment — Aggressive ischemic risk factor management
  Arms: Cardiological assessment

SUMMARY:
This is a prospective, exploratory, randomised clinical trial. Patients with diagnosed cancer that are to be treated with 5-fluorouracil (5-FU) will be randomised into standard oncological treatment or a cardiological assessment prior to the 5-FU treatment. The investigators hypothesize that aggressive management of ischemic risk factors in asymptomatic patients will reduce the number of hospitalisations and investigations for acute coronary syndrome during and after 5-FU treatment and that patients with high coronary artery calcium scores are more likely to experience chest pain during the treatment with 5-FU.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified cancer
* First-time treatment with 5-FU/Capecitabine
* Expected remaining lifetime > 6 months
* Informed consent

Exclusion Criteria:

* Known ischemic heart disease
* Ischemia-suspicious symptoms prior to 5-FU treatment
* Ischemia-suspicious ECG-changes prior to 5-FU treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Acute coronary syndrome | 6 months
  Composite endpoint of the incidence of overall mortality, chest pain requiring hospital admittance, the incidence of coronary angiography intervention and acute coronary syndrome

SECONDARY OUTCOMES:
Chest pain | 6 months
  Incidence of chest pain

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke B Hansen, MD, PhD, Principal Investigator — Vejle Hospital; Lars H Jensen, MD, PhD, Study Chair — Department of Oncology, Vejle Hospital, Denmark
Locations (1):
- Departments of Oncology and Medicine, Vejle Hospital, Vejle, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lyhne JD, Hansen VB, Vestergaard LD, Hosbond SE, Busk M, Gnanaganesh M, Maae E, Havelund BM, Hansen TF, Timm S, Jensen LH, Lyhne MD. Primary prevention of cardiotoxicity in cancer patients treated with fluoropyrimidines: a randomized controlled trial. Cardiooncology. 2025 May 17;11(1):48. doi: 10.1186/s40959-025-00344-3. PMID 40382663